CLINICAL TRIAL: NCT04552314
Title: Predictive Value of Postoperative Filtering Bleb Vascularity in Mitomycin-C Augmented Trabeculectomy
Brief Title: Bleb Vascularity and the Outcomes After Trabeculectomy
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: KE-0254/203/2014
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2020-09

CONDITIONS: Glaucoma; Filtering Bleb
Keywords: filtering bleb; trabeculectomy; glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients after primary MMC-augmented trabeculectomy

SUMMARY:
1. Study objective: To evaluate the relationship between filtering bleb vascularity and the surgical outcomes after trabeculectomy
2. Study design: A prospective study of 51 eyes of 44 patients after primary MMC-augmented trabeculectomy. The follow-up was 12 months.

DETAILED DESCRIPTION:
Total vessel area of a filtering bleb was measured with ImageJ software on colour photographs of a filtering bleb on day 1, 14, 1, 3 and 6 months and 1 year after trabeculectomy. Blebs were classified clinically as successful (IOP below 18 mmHg and a >30% reduction in IOP without antiglaucoma medications or additional surgical interventions) or failed. Linear regression analysis was performed to determine the correlation of the bleb vascularity with IOP.

ELIGIBILITY:
Inclusion Criteria:

* primary open angle glaucoma (POAG) with medically uncontrolled intraocular pressure (IOP)
* pseudoexfoliation glaucoma (PEXG) with medically uncontrolled intraocular pressure (IOP)

Exclusion Criteria:

* primary angle closure glaucoma (PACG)
* secondary glaucoma except PEXG
* previous eye surgery
* subjects with decreased vision due to other reasons than glaucoma (e.g., exudative age-related macular degeneration (AMD), proliferative diabetic retinopathy, inflammatory eye diseases)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with medically uncontrolled glaucoma who underwent primary trabeculectomy with mitomycin C (MMC) in the Department of Diagnostics and Microsurgery of Glaucoma of Medical University of Lublin, Poland
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rates of surgical success | 1 year
  The successful bleb group consisted of eyes with IOP below 18 mmHg and a >30% reduction in IOP at 1 year after surgery without antiglaucoma medications or additional surgical interventions. Failed blebs were defined when IOP was over 18 mmHg, below 18 mmHg with antiglaucoma medications or if any additional surgical intervention was necessary

SECONDARY OUTCOMES:
Correlation of Bleb vascularity with IOP | 6 months
  Linear regression analysis was performed to determine the correlation of the bleb vascularity with IOP

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Żarnowski, MD, PhD, Professor, Study Chair — Medical University in Lublin